CLINICAL TRIAL: NCT00973258
Title: Randomized Controlled Trial of Community-based Nutritional, Physical and Cognitive Training Intervention Programmes for At Risk Frail Elderly
Acronym: FIT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Medical Research Council (NMRC), Singapore (Other Government)
Collaborators: National University of Singapore (Other); Alexandra Hospital (Other); St Luke's Hospital, Singapore (Other)
Responsible Party: Principal Investigator, Ng Tze Pin, Associated professorial fellow, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NMRC/1108/2007
Record Dates: First submitted 2009-09-08; First posted 2009-09-09 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Pre-Frail or Frail State
MeSH Terms: interventions — Calcium Carbonate; Exercise; Resistance Training; Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Nutritional Intervention (Experimental): Nutritional intervention
  Interventions: Dietary Supplement: Nutritional Intervention
- Physical Exercise (Experimental): Physical exercise training intervention
  Interventions: Other: Physical Exercise
- Cognitive Training (Experimental): Cognitive training intervention
  Interventions: Other: Cognitive Training
- Combined (Experimental): Nutritional Intervention + Physical Exercise + Cognitive Training
  Interventions: Other: Combined
- Control Group (Placebo Comparator): Participants will receive their usual diet and placeboes.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Nutritional Intervention — Each subject in the nutritional intervention group is provided with a commercial liquid formula (Fortisip Multi Fibre, Nutricia), which should be taken every evening for a period of 24 weeks. Subjects are also given one capsule of iron and folate supplement (Sangobion, Merck; consisting of 1 mg folate and 29mg iron), one capsule of Vitamin B6 and vitamin B12 supplement (Neuroforte; consisting of 200mcg B12 and 200mg vit B6) and one tablet of Caltrate with Vitamin D (consisting of 200 IU vitamin D and 600 mg of calcium) for a duration of 24 weeks.
  Other Names: Fortisip; Sangobion; Neuroforte; Caltrate
  Arms: Nutritional Intervention
Other: Physical Exercise — The exercise intervention group comprises a combination of 2 types of exercise: resistance exercise and in-balance exercise. Key components in both programs are balance and strength, because these are the most prominent domains that should be addressed in at risk frail elderly. The first program is administered in the first 6-week, and then followed by the second program for the next 6-week of intervention period. Both exercise programmes are tailored to the functional needs of the participants, maintaining a moderate intensity that focuses on long-term sustainability and enjoyment.
  Other Names: Resistance exercise; In-balance exercise
  Arms: Physical Exercise
Other: Cognitive Training — The proposed cognitive training intervention program comprises:
  1. Reasoning training focusing on inductive reasoning, the ability to solve problems that follow a serial pattern and manifest in executive functioning.
  2. Memory training focusing on verbal episodic memory, which deals with acquisition and retrieval of information acquired in a particular place at a particular time.
  3. Speed training focusing on visual search and the ability to identify and locate visual information quickly in a divided attention format, with and without distractors.
  Other Names: Reasoning training; Memory training; Speed training
  Arms: Cognitive Training
Other: Combined — Nutritional Intervention + Physical Exercise + Cognitive Training
  Arms: Combined
Other: Placebo — Participants will receive their usual diet and placeboes.
  Arms: Control Group

SUMMARY:
The aims of this proposed community-based randomized controlled trial are to evaluate the effectiveness of nutritional, physical exercise and cognitive training interventions for at-risk and frail elderly, to elucidate the biological determinants and changes associated with frailty, and to develop, evaluate and demonstrate the feasibility of screening instruments for frailty.

DETAILED DESCRIPTION:
Community-living elderly persons are screened and 250 participants satisfying rigorous criteria for frailty are randomized to received nutritional, physical training, cognitive training, combined or control arms for 24 weeks and followed up for 12 months. Baseline evaluations will include an extensive range of potential markers of frailty and outcome measures, including functional disability and hospitalizations.

Frail subjects who were selected for the interventional trial (N=250) are followed up at 3, 6 and 12 months after baseline assessment. Non-trial subjects (about 2750) are followed up at 1 year after baseline assessment

ELIGIBILITY:
Inclusion Criteria:

1. Age of 65 years or older
2. Living at home
3. Able to walk without personal assistance and no other physical limitations that can limit participation and adherence, particularly to exercise intervention programme
4. Meet criteria for frailty

Operational definition of frailty.

The participants are assessed and classified on the level of frailty by the following measures and criteria:

1. Weight loss
2. Slowness
3. Poor balance and weakness assessed by chair stand test
4. Muscle weakness assessed by hand grip and knee extension strength
5. Exhaustion, fatigue or low endurance
6. Low physical activity

Exclusion Criteria:

1. Member of household already enrolled
2. Dementia or cognitive impairment, major depression or other psychotic disorders
3. Severe audio-visual impairment
4. Progressive, degenerative neurologic disease like Parkinsonism, fits/ epilepsy, etc
5. Rapidly progressive or terminal illness under palliative care with life expectancy less than 12 months
6. History of alcohol abuse or any other substance abuse
7. Severely affect muscle/joint dysfunction resulting in disability
8. Hospital admission in the past 3 months
9. Regular physical training or physiotherapy or current participation in a vigorous exercise or weight-training program more than once per week
10. Undergoing therapeutic diet incompatible with nutritional supplementation
11. In the opinion of research clinician, the intervention is deemed to be potentially hazardous for the subject, such as serious cardiac and pulmonary disease.

Ages: 65 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 246 (Actual)
Dates: Start 2009-12; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Reduction of frailty | 12 months
Frailty score (continuous variable) | 12 months
Measures of frailty components (BMI, fast gait speed test, knee extension, exhaustion score and time spent on physical activities per day). | 12 months

SECONDARY OUTCOMES:
Frequency of falls (defined as an event resulting in a person coming to rest unintentionally on the ground or other lower level; near-falls are not included; Robertson, 2001). | 12 months
Health service utilization (frequencies of doctor visits, emergency room visit, hospitalization, nursing home admission) | 12 months
Mortality | 12 months
Disability in activities of daily living (ADL) and instrumental activities of daily living (IADL). | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Tze-Pin Ng, MD, Principal Investigator — National University of Singapore
Locations (1):
- Alexandra Hospital, Singapore, Singapore, Singapore

REFERENCES:
- [Derived] Ng TP, Feng L, Nyunt MS, Feng L, Niti M, Tan BY, Chan G, Khoo SA, Chan SM, Yap P, Yap KB. Nutritional, Physical, Cognitive, and Combination Interventions and Frailty Reversal Among Older Adults: A Randomized Controlled Trial. Am J Med. 2015 Nov;128(11):1225-1236.e1. doi: 10.1016/j.amjmed.2015.06.017. Epub 2015 Jul 6. PMID 26159634